CLINICAL TRIAL: NCT03599219
Title: Prevalence of Platelet Dysfunction Inblood With a Bleeding History
Brief Title: Platelet Dysfunction in Blood Donors
Acronym: DysPlaq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etablissement Français du Sang (Other)
Collaborators: University of Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APR2016-27; 2016-A00117-44 (Registry Identifier: RCB)
Record Dates: First submitted 2018-02-27; First posted 2018-07-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Platelet Dysfunction in Blood Donors
Keywords: platelets; bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: prospective case control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Other): donors with an hemorrhagic score >2 and / or hematoma (more than 4 cm) that occurred during blood donation
  Interventions: Biological: sample
- control (Other): donors with an hemorrhagic score <2.
  Interventions: Biological: sample

INTERVENTIONS:
Biological: sample — confirmation of platelet dysfunction
  Other Names: questionnary to obtain an hemorrhagic score

SUMMARY:
Platelets are circulating blood cells. They bind to each other and to the damaged vessel wall to prevent excessive bllod loss. Unlike quantitative platelet defects, there is no automated, simple test to diagnose qualitative platelets defects. However, these defects expose to bleeding in a surgical situation and could explain the transfusion inefficiency of some platelet concentrates.

In recent decades, considerable progress has been made in understanding qualitative platelet disorders.

In this project, we propose to submit blood donors to a standardized hemorrhagic diathesis questionnaire and to compare the prevalence of platelet function abnormalities in blood donors with and without hemorrhagic diathesis.

DETAILED DESCRIPTION:
Primary objective specify the prevalence of qualitative platelet disorders in blood donors with i) a clinical history of bleeding diathesis collected through a standardized and validated questionnaire ii) and / or a hematoma (more than 4 cm) that occurred during blood donation.

Secondary objectives to obtain the prevalence of other defects of hemostasis

ELIGIBILITY:
Inclusion Criteria:

- Any male or female volunteer eligible for the blood donation

Exclusion Criteria:

* Subject with contraindications to blood donation:
* weight <50 kg;
* severe fatigue,
* anemia,
* insulin-dependent diabetes;
* subject treated for epileptic seizures or having followed a treatment whose arrest is less than 14 days old.
* active pregnancy or childbirth less than 6 months old.
* viral disease (eg influenza, gastroenteritis ...) active less than two weeks after the end of symptoms.
* waiting period not respected after certain acts of daily life according to the regulatory criteria set by the EFS
* HIV infection, hepatitis B, hepatitis C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Platelet functions | first visit 1 week
  Quantification of surface platelet proteins by flow cytometry

SECONDARY OUTCOMES:
Exploration of Coagulation | first visit 1 week
  Von Willebrand factor quantification

CONTACTS AND LOCATIONS:
Overall Officials: Picard Christophe, Dr, Principal Investigator — Etablissement francais du sang
Locations (1):
- Maison Du Don, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided